CLINICAL TRIAL: NCT00170859
Title: A One-year Multicenter, Randomized, Open-label Study of the Safety and Efficacy of Everolimus Versus Mycophenolate Mofetil in Combination With Reduced Dose Cyclosporine Microemulsion in Maintenance Heart Transplant Recipients
Brief Title: Everolimus Versus Mycophenolate Mofetil in Combination With Reduced Dose Cyclosporine Microemulsion in Maintenance Heart Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001ADE01
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Heart Transplantation
Keywords: everolimus; cyclosporine microemulsion; renal function
MeSH Terms: interventions — Everolimus

INTERVENTIONS:
Drug: Everolimus

SUMMARY:
In this study two immunosuppressive regimens (everolimus in combination with cyclosporine microemulsion and mycophenolate mofetil with cyclosporine microemulsion) with reduced dose cyclosporine microemulsion are compared in maintenance heart transplant recipients with impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of primary heart transplant
* Reduced renal function (serum creatinine > 1.7 ng/mL over 2 months or more) at 6 months or more after heart transplantation
* Patients with current immunosuppressive therapy consisting of cyclosporine microemulsion and mycophenolate mofetil

Exclusion Criteria:

* Patients who are recipients of multiple organ transplants
* Patients who have previously received an organ transplant
* Patients with serum creatinine > 3.5 mg/dl

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-08; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigational Site, Various Cities, Germany

REFERENCES:
- [Result] Bara C, Dengler T, Hack MA, Ladenburger S, Lehmkuhl HB. A 1-year randomized controlled study of everolimus versus mycophenolate mofetil with reduced-dose cyclosporine in maintenance heart transplant recipients. Transplant Proc. 2013 Jul-Aug;45(6):2387-92. doi: 10.1016/j.transproceed.2013.03.032. PMID 23953553